CLINICAL TRIAL: NCT04488146
Title: Epidemiology and Characterization of Pain in Patients With Crohn Disease
Brief Title: Pain in Patients With Crohn Disease (PAINCD)
Acronym: PAINCD
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Liege (Other)
Responsible Party: Principal Investigator, Jean François Brichant, Professor of Anesthesiology, University of Liege
Other Study IDs: PAINCD
Record Dates: First submitted 2020-07-15; First posted 2020-07-27 (Actual); Last update posted 2020-07-27 (Actual); Status verified 2020-07

CONDITIONS: Crohn Disease; Pain; Depression, Anxiety
Keywords: crohn disease; pain
MeSH Terms: conditions — Crohn Disease; Pain; Depression; Anxiety Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Abdominal pain is a common symptom in patients with Crohn disease (CD). Pain is multifactorial, may result from inflammation but persists in many patients during remission.

The aim of our study is to determine the epidemiology of pain in CD patients and define the characteristics of pain : localisation, temporal and sensorial characteristics, neuropathic component, impact on quality of life and mood.

DETAILED DESCRIPTION:
Abdominal pain is a common symptom in patients with inflammatory bowel disease (IBD) that alters quality of life and can lead to increased healthcare utilization. In addition to abdominal pain, pain can result from extra-intestinal manifestation of IBD. 40% of IBD patients suffer from extra-intestinal manifestations. Although abdominal pain has been traditionally attributed to inflammation, functional abdominal pain exists in patients with IBD, associated with a variety of potential causes. About 20-40% of patients in complete clinical and endoscopic remission continue to experience chronic pain. Thus, when examining an IBD patient with abdominal pain, in addition to IBD-related complications (e.g., inflammation, stricture), it is important to screen for other contributors, including peripheral factors (visceral hypersensitivity, bacterial overgrowth, and bowel dysmotility) and centrally mediated neurobiological and psychosocial underpinnings. These central factors include psychological symptoms, sleep disturbance, and stress. Opioid-induced hyperalgesia (e.g., narcotic bowel syndrome) is also growing in recognition as a potential central source of abdominal pain.

Pronounced severe pain impacts health related quality of life (QoL). Longstanding pain leads to decreased QoL, increase in pain medication intake, and co-morbidities including depression, anxiety and even addiction. Furthermore, pain attacks severely interfere with social and professional life.

Knowledge of these potential aetiologies should be used to individualize treatment of abdominal pain in patients with IBD. Accurate assessment of the source of pain can help guide appropriate diagnosis workup and use of modifying therapy.

The aim of the study is to determine the epidemiology of pain in patients with Crohn disease (CD) and to characterize their pain (localisation, temporal characteristics, acute vs. chronic, sensorial characteristics, existence of neuropathic component, existence of hyperalgesia), and their impact of QoL, depression and anxiety

ELIGIBILITY:
Inclusion Criteria:

* any patient with Crohn disease in remission or relapse period age ≥ 18 yo.

Exclusion Criteria:

* No exclusion criteria beside no informed consent and inadequate French language skills

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any patient visiting the multidisciplinary center for inflammatory bowel diseaese chaired by Prof Edouard Louis at CHU Liège, domaine du Sart Tilman, Liège, Belgium
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-10 (Estimated); Primary Completion 2021-01 (Estimated); Study Completion 2021-02 (Estimated)

PRIMARY OUTCOMES:
Pain intensity in patients with Crohn Disease (CD) | During the last 30 days
  Pain intensity measured using a 100 mm visual analog scale (0 = no pain; 100 the worst imaginable pain)

SECONDARY OUTCOMES:
Presence of hyperalgesia | During the last 30 days
  Using Von Frey hairs (size 2.83 for dectection of allodynia; size 6.65 for temporal somation)
Search for a neuropathic component of pain | During the last 30 days
  Using DN-4 questionnaires : a score ≥ 3 = neuropathic component
Investigation of the impact of pain on depression and anxietey | During the last 30 days
  Using the HAD (Hospital anxiety depression) scale : as score > 11 = true symptomatology

CONTACTS AND LOCATIONS:
Overall Officials: Jean-François Brichant, M.D., Principal Investigator — CHU Liege, Domaine du Sart Tilman, Liege, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Srinath A, Young E, Szigethy E. Pain management in patients with inflammatory bowel disease: translational approaches from bench to bedside. Inflamm Bowel Dis. 2014 Dec;20(12):2433-49. doi: 10.1097/MIB.0000000000000170. PMID 25208108
- [Result] Morrison G, Van Langenberg DR, Gibson SJ, Gibson PR. Chronic pain in inflammatory bowel disease: characteristics and associations of a hospital-based cohort. Inflamm Bowel Dis. 2013 May;19(6):1210-7. doi: 10.1097/MIB.0b013e318280e729. PMID 23524595
- [Result] Zeitz J, Ak M, Muller-Mottet S, Scharl S, Biedermann L, Fournier N, Frei P, Pittet V, Scharl M, Fried M, Rogler G, Vavricka S; Swiss IBD Cohort Study Group. Pain in IBD Patients: Very Frequent and Frequently Insufficiently Taken into Account. PLoS One. 2016 Jun 22;11(6):e0156666. doi: 10.1371/journal.pone.0156666. eCollection 2016. PMID 27332879
- [Derived] Hardy PY, Fikri J, Libbrecht D, Louis E, Joris J. Pain Characteristics in Patients with Inflammatory Bowel Disease: A Monocentric Cross-Sectional Study. J Crohns Colitis. 2022 Sep 8;16(9):1363-1371. doi: 10.1093/ecco-jcc/jjac051. PMID 35380673